CLINICAL TRIAL: NCT03655054
Title: SUBCUTANEOUS TIBIAL NERVE STIMULATION FOR URGENCY URINARY INCONTINENCE: A FOLLOW-ON STUDY
Brief Title: eCoin for OAB Feasibility Follow-on Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Valencia Technologies Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 111-3335
Record Dates: First submitted 2018-08-29; First posted 2018-08-31 (Actual); Results first posted 2021-04-26 (Actual); Last update posted 2022-10-17 (Actual); Status verified 2022-10

CONDITIONS: Overactive Bladder; Urge Incontinence; Incontinence, Urinary; Urinary Urge Incontinence
MeSH Terms: conditions — Urinary Bladder, Overactive; Urinary Incontinence, Urge; Urinary Incontinence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- eCoin Tibial Nerve Stimulation (Experimental)
  Interventions: Device: eCoin Tibial Nerve Stimulation

INTERVENTIONS:
Device: eCoin Tibial Nerve Stimulation — Subcutaneous stimulation of the tibial nerve using the eCoin device.

SUMMARY:
This trial is a prospective, multicenter, single-arm follow-on study will evaluate the safety and effectiveness of eCoinTM tibial nerve stimulation in subjects with urgency urinary incontinence (UUI) as defined by the American Urological Association (30). The follow-on study will evaluate changes from baseline in OAB symptoms as measured by voiding diaries and patient-reported outcomes through 24 weeks of eCoinTM therapy (which is the same as 28 weeks from study device reimplantation).

ELIGIBILITY:
Inclusion Criteria:

1. Individual participated in the eCoin Feasibility Study for Urgency Urinary Incontinence.
2. Individual was implanted with the study device during the eCoin Feasibility Study for Urgency Urinary Incontinence.

Exclusion Criteria:

1. In the opinion of the investigator, individual is not a good candidate for participation in the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2019-03-13 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2022-09-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (7):
- United States (4):
  - The Clark Center for Urogynecology, Newport Beach, California
  - UnityPoint Clinic, Waterloo, Iowa
  - Alliance Urology Specialists, Greensboro, North Carolina
  - The Institute for Female Pelvic Medicine & Reconstructive Surgery (FPM Institute), Allentown, Pennsylvania
- New Zealand (3):
  - Urology Associates, Christchurch
  - Roundhay Medical Centre, Nelson
  - Tauranga Urology Research Ltd, Tauranga

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kaaki B, English S, Gilling P, Meffan P, Lucente V, MacDiarmid S, Clark M, Sen SK. Six-Month Outcomes of Reimplantation of a Coin-Sized Tibial Nerve Stimulator for the Treatment of Overactive Bladder Syndrome With Urgency Urinary Incontinence. Female Pelvic Med Reconstr Surg. 2022 May 1;28(5):287-292. doi: 10.1097/SPV.0000000000001105. Epub 2022 Sep 22. PMID 35536667

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | eCoin Tibial Nerve Stimulation
Started | 23
Completed | 22
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | eCoin Tibial Nerve Stimulation
Number analyzed (Participants) | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.6 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 23
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 23
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  New Zealand | 9
  United States | 14
Mean UUI Episodes/Day [Mean (Standard Deviation); unit: episodes/day] | 4.8 (3.2)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Urgency Urinary Incontinence Episodes as Measured by a 3-day Voiding Diary.
Time Frame: 12 weeks after device activation.
Measure: Mean (Standard Deviation); unit: episodes/day
Arm/Group | eCoin Tibial Nerve Stimulation
Number analyzed (Participants) | 23
episodes/day | -2.2 (3.3)

2. Primary Outcome: Safety in All Patients. All Adverse Events Will be Reported in All Patients Who Were Implanted 4 Months After Implantation.
Description: Instances of a related adverse event.
Time Frame: 16 weeks after device implantation.
Measure: Number; unit: adverse events
Arm/Group | eCoin Tibial Nerve Stimulation
Number analyzed (Participants) | 23
adverse events | 8

3. Secondary Outcome: Change From Baseline in Urgency Urinary Incontinence Episodes as Measured by a 3-day Voiding Diary.
Time Frame: 24 weeks after device activation.
Measure: Mean (Standard Deviation); unit: episodes/day
Arm/Group | eCoin Tibial Nerve Stimulation
Number analyzed (Participants) | 22
episodes/day | -3.7 (1.2)

4. Secondary Outcome: Safety in All Patients. All Adverse Events Will be Reported in All Patients Who Were Implanted 6 Months After Implantation.
Description: Instances of a related adverse event
Time Frame: 28 weeks after device implantation.
Measure: Number; unit: adverse events
Arm/Group | eCoin Tibial Nerve Stimulation
Number analyzed (Participants) | 22
adverse events | 8

ADVERSE EVENTS:
Time Frame: 28 weeks after implantation
Arm/Group | eCoin Tibial Nerve Stimulation
All-Cause Mortality (participants affected / at risk) | 0/23
Serious Adverse Events (participants affected / at risk) | 0/23
Other Adverse Events (participants affected / at risk) | 6/23
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | eCoin Tibial Nerve Stimulation (N=23)
Incision site erythema (Skin and subcutaneous tissue disorders) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1)
Incision site discomfort (General disorders) | 3 (3)
Incision site swelling (General disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-13): https://cdn.clinicaltrials.gov/large-docs/54/NCT03655054/Prot_SAP_000.pdf